CLINICAL TRIAL: NCT05373537
Title: Pilot RCT to Compare a Home Based Tailored Cognitive Behavioral Therapy for Insomnia (CBT-I) Versus Webased CBT-I to Improve Sleep in Caregivers With Insomnia in the Context of Caring for a Child With Autism Spectrum Disorder
Brief Title: Treatment to Improve Sleep in Caregivers With Insomnia and a Child With Autism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 850797
Record Dates: First submitted 2022-04-11; First posted 2022-05-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Insomnia Chronic; Caregiver Burden
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders; Caregiver Burden | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Pilot Randomized control trial Comparing a home-based vs a web-based approach to CBT-Insomnia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based (Experimental): home- based CBT-Insomnia intervention
  Interventions: Behavioral: Cognitive behavioral therapy for Insomnia
- web-based (Experimental): web-based CBT-Insomnia intervention
  Interventions: Behavioral: Cognitive behavioral therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for Insomnia — Caregiver with insomnia will receive CBT-Insomnia and will be trained to implement CBT-I tailored for their child with Autism Spectrum Disorder and Insomnia

SUMMARY:
Autism Spectrum Disorder (ASD) represents one of the most perplexing neurobiological disorders with a prevalence of 1 in 54 children. The lifelong challenging and disruptive behaviors often associated with ASD requires caregivers to change their behavior and modify their environments to provide an ecosystem for optimal outcomes for their child, family and themselves. ASD behaviors can have significant impact on caregivers mental health and family functioning, including the ability to develop and maintain healthy sleep routines. The caregiving population in US has a high prevalence of insomnia; two thirds of caregivers experiencing difficulties falling and/or staying asleep. The prevalence of insomnia in children with ASD is equally high, 60-80% experiencing night waking contributing to poor daytime behavior and disrupted sleep in the caregivers. This pilot RCT will focus on improving caregivers sleep in the context of caring for a child with ASD and insomnia with a multi-disciplinary team. The investigators will compare a home-based tailored CBT for Insomnia (CBT-I) versus a web-based Way to Health CBT-I intervention. This data will support a larger RCT with the Department of Defense funding opportunity through the Congressionally Directed Medical Research Program. This Autism Research Program focuses on improving lives of those living with ASD.

DETAILED DESCRIPTION:
Overall objectives

The investigators propose to compare a home-based tailored CBT-I intervention versus a web-based Way to Health (WTH) platform tailored CBT-I intervention for caregivers with insomnia in the context of caring for a child with ASD and insomnia. This pilot RCT will further the investigators previous work and investigate the feasibility, acceptability, and efficacy of a web based versus home-based CBT-I intervention for both the caregiver with insomnia and the child with ASD and insomnia. The investigators also hope to gain a greater understanding of the relationships between child and caregiver sleep, caregiver psychiatric conditions, child behavior, and maternal self-efficacy. These findings will provide preliminary data for a larger RCT to improve sleep for all family members. The specific aims of this pilot study are:

1. To determine the acceptability and feasibility of a RCT design utilizing a novel, web-based WTH platform versus a home- based CBT-I intervention to improve sleep of a caregiver with insomnia and a child with ASD and insomnia. The investigators plan to evaluate the recruitment, retention, randomization, and training required for this study.
2. To examine the relationship between caregiver self- efficacy, caregiver psychiatric conditions and sleep, and child daytime behaviors and sleep pre and post intervention.
3. To compare the effect of a home- based tailored CBT-I versus web based WTH CBT-I on child and caregiver sleep with a primary endpoint of total sleep time and sleep latency measured with Actigraphy, caregiver mental health scores, and child daytime behaviors.

Primary outcome variable(s)

1. To determine the acceptability and feasibility of a RCT design with the Opinion Survey assessing acceptability with an 8 items rated on a 7- point Likert scale survey This study will be considered feasible if we obtain a 70% completion rate for the repeated measures. Acceptability of the web-based and home based will be determined by parent acceptability survey. This protocol will be considered acceptable to parents if the acceptability score is 70% or greater.
2. To compare the effect of a home- based tailored CBT-I versus web based WTH CBT-I on child and caregiver sleep with a primary endpoint of total sleep time and sleep latency measured with Actigraphy Secondary outcome variable(s) To examine the relationship between caregiver self- efficacy, caregiver psychiatric conditions, child daytime behaviors and sleep parameters pre and post intervention. To examine the mediation effect of caregiver self-efficacy on the relationship between depressive symptoms, caregiver and child sleep, and child symptom severity and behavior, the investigators will use the Baron and Kenny 4-step regression model.71 Independent predictors of depressive symptoms will be tested and adjusted in all analytical steps. Mediation analysis will be performed for all subjects in a pooled sample, followed by a sensitivity analysis to determine the moderating role of child's symptom severity. Conduct a Sobel test to analyze the statistical significance of the mediation effect.

Background Autism Spectrum Disorder (ASD) represents one of the most perplexing neurobiological disorders with a prevalence of 1 in 54 children (1). Substantial heterogeneity exists in the degree of impairment, the collection of behavioral symptoms and the medical conditions associated with ASD. The lifelong challenging and disruptive behaviors often associated with ASD require caregivers to change their behavior and modify their environments to provide an ecosystem for optimal outcomes for their child, family and themselves. However, ASD behaviors can have a significant impact on caregivers mental health and family functioning, including the ability to develop and maintain healthy sleep routines (2). The caregiving population in the U.S. has a high prevalence of insomnia, with two thirds of caregivers experiencing difficulties falling and/or staying asleep. The prevalence of insomnia in children with ASD is equally high, with 60-80% experiencing night waking, contributing to poor daytime child behavior and disrupted caregiver sleep (3, 4). This pilot RCT will focus on improving caregivers sleep in the context of caring for a child with ASD and insomnia with a multi-disciplinary team approach. This pilot data will support a larger RCT with the Department of Defense (DoD) funding opportunity through the Congressionally Directed Medical Research Program. This Autism Research Program focuses on improving lives of those living with ASD.

The investigators recently completed study reveals that 36.6 % of mothers of children with ASD report a psychiatric disorder before and during pregnancy (5). Moreover, 30% of mothers of children with ASD report depression (6-13), revealing the significant vulnerability of this caregiving population. Evidence suggests that insomnia can be a precursor to onset or worsening of psychiatric conditions (14). Maternal depression is associated with lower family functioning, which affects physical, behavioral, and emotional outcomes of children (15-18). Notably, mothers depressive symptoms can interfere with and even blunt the effects of home-based interventions for children with ASD (8). This results in a cycle of poor child outcomes and greater need for intervention (19, 20). Our study of mothers of children with ASD demonstrated that maternal depression and self-efficacy impact child behaviors (21). Therefore, the investigators hypothesize that helping caregivers improve their sleep and their childs sleep, will have a positive impact on mood, cognition, and maternal self-efficacy. Yet, little is known about how family interventions may improve sleep behaviors and mental health in this vulnerable population.

The investigators previously completed RCT examined a home based, modified Cognitive Behavioral Therapy for Insomnia (CBT-I) intervention for children with ASD and insomnia (3, 4). The modified CBT-I is an 8 week intervention developed by the Principal Investigator that includes 1) A one hour education session developed by the Autism Treatment Network, Sleep Tool Kit (Appendix A); 2) Identifying positive evening routines, developing a visual schedule and implementing ecological changes to the bedroom, 3) Introducing a calming module with a choice of 5-12 soothing activities selected by the caregiver/child (Appendix B); and 3) Developing a bedtime protocol pairing irresistible sleepiness with the bedroom (stimulus control). The investigators study, using actigraphy an objective measure of sleep, showed that tailored CBT-I (n=20) decreased wake time in bed by 65 minutes with an effect size=1.05 compared to 19 minutes with an effect size=0.26 in the sleep education only group (n=16). The investigators study suggested that the tailored CBT-I has a larger effect than sleep education on sleep in children with ASD. However, this intervention required frequent and costly home visits by a multi-disciplinary team. In addition, 40% of mothers expressed that they had difficulty implementing CBT-I for their children due to exhaustion and feelings of being overwhelmed related to their own mental health.

To address this gap, the investigators propose to compare a home-based tailored CBT-I intervention versus a web-based Way to Health (WTH) platform tailored CBT-I intervention for caregivers with insomnia in the context of caring for a child with ASD and insomnia. This pilot RCT will further previous work and investigate the feasibility, acceptability, and efficacy of a web based versus home-based CBT-I intervention for both the caregiver with insomnia and the child with ASD and insomnia. The investigators also hope to gain a greater understanding of the relationships between child and caregiver sleep, caregiver psychiatric conditions, child behavior, and maternal self-efficacy. These findings will provide preliminary data for a larger RCT to improve sleep for all family members.

ELIGIBILITY:
Inclusion Criteria for Caregiver with a child with ASD:

* Caregiver age 18 years or older
* Diagnosis of Insomnia
* Parental/guardian will give permission (informed consent) for child
* Telephone and web Access
* Stable medical and behavioral conditions, with no change in health status in the past three months
* Commitment to maintaining stable medication doses and keeping medication consistent

Inclusion Criteria for Children with ASD:

* Children age 3 to 17 years and one of their parents
* Diagnosis of Autism Spectrum Disorders, confirmed with Autism Diagnostic Observation Schedule and/or DSM-IV criteria.
* Diagnosis of Behavioral Insomnia or Insomnia due to ASD (Insomnia due to internal
* Parental/guardian permission (informed consent) and if appropriate, child assent.
* Telephone and web Access
* Stable medical and behavioral conditions, with no change in health status in the past
* Commitment to maintaining stable medication doses and keeping child's sleep medication consistent

Key exclusion criteria for Caregiver and child with ASD:

* Insomnia due to co-occurring medical conditions and/ or sleep disorders such as obstructive sleep apnea (OSA), narcolepsy, restless leg syndrome, severe reflux, nocturnal asthma
* Unstable co-occurring medical conditions such as epilepsy or other neurological disorders, sickle cell anemia, diabetes or severe eczema
* Significant hearing or vision loss
* Known genetic disorders such as Fragile X, 22ql 1.2 Deletion Syndrome, Rett Disorder, Down Syndrome.
* Subjects who, in the opinion of the Investigator, may be non¬ compliant with study schedules or procedures.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Caregiver Acceptability Opinion Survey | At week 8
  Opinion Survey with 8 items rated on a 7- point Likert scale. minimum of 0 and max of 56 with a score of 40 or greater will be considered acceptable for this study.
Feasibility of pilot study | At week 8
  This study will be considered feasible if we obtain a 70% completion rate for the all measures.

SECONDARY OUTCOMES:
Change in reported sleep on sleep diaries | 8 weeks
  Participants will be asked to record the amount of sleep each night
Change in Caregiver behaviors | week 8
  Depression questionnaire: Patient Health Questionnaire -9 with a minimum score of 0 and max of 27 with lower scores representing better outcome
Change in Child Daytime behaviors | week 8
  Child Behavior Checklist (CBCL) T scores of 0 to 100 with lower scores representing better outcome
Change in total sleep time average measured by an actigraphy watch for caregiver | week 8
  Total sleep time in minutes on average for the week
Change in sleep latency as measured by actigraphy watch for caregiver | week 8
  sleep latency in minutes on average for the week
Change in wake after sleep onset as measured by by actigraphy watch for caregiver | week 8
  wake after sleep onset in minutes on average for the week
Change in total sleep time as measured by actigraphy watch for child | week 8
  Total sleep time in minutes on average for the week
Change in sleep latency as measured by actigraphy watch for child | week 8
  sleep latency in minutes on average for the week
Change in wake after sleep onset as measured by actigraphy for child | week 8
  wake after sleep onset in minutes on average for the week
Change in Maternal Self-efficacy | week 8
  Maternal-Self efficacy Scale, 10 items with minimum score of 10 and maximum of 40 with higher scores representing better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing of all underlie results in publications
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: starting 6 months after publications
Access Criteria: The PIs will review requests for access